CLINICAL TRIAL: NCT05841342
Title: A Prospective Study of Immune Function and PD-1 Antibody Therapy Efficacy Predictors for Chronic Active Epstein-Barr Virus Infection and Epstein-Barr Virus Associated Hemophagocytic Lymphohistiocytosis
Brief Title: Prospective Study of Immune Function and PD-1 Antibody Therapy Efficacy Predictors on CAEBV and EBV-HLH Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Clinical Professor, Beijing Friendship Hospital
Other Study IDs: BFH20221009004
Record Dates: First submitted 2023-04-22; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Secondary Hemophagocytic Lymphohistiocytosis; Chronic Active Epstein-Barr Virus Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10ml venous blood was extracted and peripheral blood mononuclear cells were extracted for flow cytometry detection. The detection contents included the frequencies of lymphocyte subsets, the positive proportion of PD-1/PD-L1 and EBER positive proportion in each subgroup.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Healthy male or female aged 2-80 years with negative EBV-DNA quantitative test results within the last week.
  Interventions: Other: No intervention
- CAEBV or EBV-HLH Patients: Patients aged 2-80 years who fulfilled the diagnostic criteria for CAEBV or EBV-HLH.
  The diagnostic criteria for CAEBV as defined in the recently revised World Health Organization classification include persistent IM-like symptoms for more than three months, increased EBV DNA (>10^2.5 copies/mg) in peripheral blood, histological evidence of organ disease, and EBV RNA or viral protein in affected tissues.
  Patients diagnosed with EBV-HLH must meet five of the following eight HLH-2004 diagnostic criteria:
  1. temperature 38.5 ℃ and above;
  2. splenomegaly;
  3. two or three lines of hemocytopenia, i.e. hemoglobin (HB) <90 g/L, platelets (PLT) <100 × 10^9/L or neutrophils (N) <1 × 10^9/L;
  4. triacylglycerol (TG) ≥ 3 mmol/ L or fibrinogen (Fbg) <1.5 g/L;
  5. serum ferritin (SF) ≥ 500 mg/L;
  6. phagocytosis found in bone marrow, spleen, liver or lymph nodes;
  7. soluble CD25 (sCD25) ≥ 2400 U/mL;
  8. low or absent natural killer (NK) cell activity.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This prospective case-control study aims to evaluate the immune function and find PD-1 antibody efficacy predictors on Chronic Active Epstein-Barr Virus Infection and Epstein-Barr virus-associated hemophagocytic lymphohistiocytosis by detecting lymphocyte subsets proportions in peripheral blood mononuclear cells and the positive proportion of PD-1, PD-L1 and other indicators in each lymphocyte subsets in healthy people and patients using flow cytometry before and after the initial PD-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria of EBV-HLH or CAEBV (except B lymphocytes involvement only) after the detection of EBV lymphocyte subsets. EBV-HLH diagnostic criteria: Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria; EBV-DNA in peripheral blood or EBER in tissue were positive, patients were diagnosed with EBV associated HLH (EBV-HLH). CAEBV diagnostic criteria: (1) persistent or recurrent infectious mononucleosis-like symptoms persisting for more than 3 months; (2) EBV-DNA quantitative increase in peripheral blood or tissue lesions; (3) exclusion of other possible Diagnosis, such as primary Epstein-Barr virus infection (infectious mononucleosis), autoimmune disease, congenital immunodeficiency, human immunodeficiency virus (HIV) infection, or other underlying conditions requiring immunosuppressive therapy or underlying immunosuppression.
2. Before the start of the study, total bilirubin ≤10 times the upper limit of normal, serum creatinine ≤1.5 times the normal value; fibrinogen can be corrected to ≥0.6g/L after infusion.
3. Serum HIV antigen or antibody negative.
4. HCV antibody negative, or HCV antibody positive, but HCV RNA negative.
5. HBV surface antigen and HBV core antibody are both negative. If any of the above is positive, peripheral blood hepatitis B virus DNA titer detection is required, and the number of copies less than 1×103 copies/ml can be included in the group.
6. LVEF ≥ 50% by cardiac echocardiography.
7. Women of childbearing age must be confirmed by a pregnancy test that they are not pregnant, and are willing to take effective contraceptive measures during the test period and within ≥ 12 months after the last dose. Women during pregnancy and lactation cannot participate. Contraceptive measures should be taken during the test period and within ≥3 months after the last dose.
8. Informed consent obtained.

Exclusion Criteria:

1. According to the New York Heart Association (NYHA) score, patients with heart disease of grade II or above (including grade II);
2. Pregnant or lactating women and patients of childbearing age who refused to take appropriate contraceptive measures during this trial.
3. Those who are allergic to rituximab ingredients or have more severe allergic constitution;
4. Severe hypogammaglobulinemia.
5. Active massive hemorrhage of internal organs (including gastrointestinal hemorrhage, alveolar hemorrhage, intracranial hemorrhage, etc.);
6. Uncontrolled active infection (including lung infection, intestinal infection, etc.);
7. HBV surface antigen and/or HBV core antibody are positive, and the peripheral blood hepatitis B virus DNA test confirms the existence of active hepatitis B patients.
8. Severe mental illness;
9. Patients who were not compliant during the trial and/or follow-up period.
10. Concurrently participate in other clinical investigators.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy people and patients with CAEBV or secondary EBV-HLH.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
EBV-DNA | Change from before and 2 weeks after initiating PD-1 blockade therapy.
  Treatment effectiveness is defined: EBV-DNA copies/ml in peripheral blood turns negative, and the involved tissues (such as lymph nodes, bone marrow, skin, etc.) are negative in EBER test or the EBV copy number has decreased by more than 2 orders of magnitude, but it is still positive.

SECONDARY OUTCOMES:
CAEBV Evaluation of treatment response | Change from before and 2 weeks after initiating PD-1 blockade therapy.
  Complete response (CR) was defined as EBV-DNA copy number below the lower limit of detection (<5.0×10^2 copies/ml) for at least 4 weeks.
  Partial response (PR) was defined as ≤ 1/100 reduction in EBV-DNA copy number, and the CR criterion was not met.
  Failure to achieve at least PR was defined as no response (NR). Besides, the main clinical manifestation of CAEBV, including fever, asthenia, liver damage (elevation of ALT and AST), skin rash, cytopenia and lymphadenopathy was also evaluated.
EBV-HLH Evaluation of treatment response | Change from before and 2 weeks after initiating PD-1 blockade therapy.
  A complete response (CR) was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response (PR) was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×10^9/L, a response was defined as an increase by at least 100% to>0.5×10^9/L; for patients with a neutrophil count of 0.5 to 2.0× 109/L, an increase by at least 100% to >2.0 × 10^9/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.
Progression Free Survival | 6 months
  from date of inclusion to date of progression, relapse, or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China